CLINICAL TRIAL: NCT06764810
Title: Association Between Motor Skills and Sensory Profiles in Children With Typical and Atypical Development Aged 4 to 11 Years: A Cross-Sectional Observational Case-Control Study
Brief Title: Association Between Motor Skills and Sensory Profiles in Children With Typical and Atypical Development Aged 4 to 11 Years
Acronym: MOTISEN
Status: Recruiting | Type: Observational
Sponsor: University of Vic - Central University of Catalonia (Other)
Responsible Party: Principal Investigator, Mirari Ochandorena Acha, PhD, University of Vic - Central University of Catalonia
Other Study IDs: MOTISEN01; 006_2024 (Other Grant/Funding Number: Catalan Board of Physical Therapy)
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Developmental Disability; Autism Spectrum Disorder; Development Coordination Disorder; Attention Deficit Disorder With Hyperactivity; Typical Development
Keywords: motor skills disorders; physical therapy modalities; pediatrics; child development
MeSH Terms: conditions — Developmental Disabilities; Autism Spectrum Disorder; Motor Skills Disorders; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Typical development: Children aged 4 to 11 years will be recruited from the local community, including schools and social networks connected to the research team.
  Recruitment will follow the same protocol as for the atypical cohort, including the use of an information sheet and video link to explain the study's aims, methodology, and voluntary participation.
  Inclusion Criteria:
  Children aged 4 to 11 years with no history or diagnosis of developmental, neurological, or sensory disorders.
  Reported by parents as meeting typical developmental milestones.
  Exclusion Criteria:
  Children with reported or observed delays in motor or sensory development. Presence of medical conditions (e.g., chronic illness, vision or hearing impairments) that could affect sensory or motor performance.
  Data on age, gender, gestational history, birth weight, family type (e.g., nuclear, single-parent), and parents' educational levels will be collected to characterize the cohort.
- Atypical development: Children aged 4 to 11 years with atypical neurodevelopment (ASD, ADHD, DCD) will be recruited from CDIAP Tris Tras, Neuro Xics, and Criv in Vic.
  Parents will receive an information sheet and video explaining the study objectives, methods, and participation requirements.
  Inclusion Criteria:
  Diagnosed or reported atypical neurodevelopment:
  ASD: Subclinical symptoms or Level 1 diagnosis. ADHD: Predominantly inattentive, hyperactive/impulsive, or combined presentation; children under six exhibiting typical ADHD behaviors.
  DCD: Diagnosed or meeting criteria for motor skills below age expectations, impacting daily life or school performance, and not explained by another condition.
  Aged 4 to 11 years. Parent/legal guardian consent.
  Exclusion Criteria:
  Moderate to severe intellectual disability (IQ ≤ 51) neurological disorders, severe behavioral/mental health issues, or sensory impairments affecting motor/sensory assessments.

SUMMARY:
Background and Justification Childhood developmental disorders, such as Autism Spectrum Disorder (ASD), Attention Deficit Hyperactivity Disorder (ADHD), and Developmental Coordination Disorder (DCD), pose significant challenges for children and their families. These disorders impact children's growth and learning, leading to difficulties in key areas such as language, communication, behavior, social interaction, and motor skills. Research in this area is limited, particularly regarding fine and gross motor skills in relation to sensory processing in children with these diagnoses.

Hypothesis and Objectives There is an association between motor skills and sensory processing in children aged 4 to 11 years, depending on whether they have typical or atypical neurodevelopment, such as ASD, ADHD, and DCD.

Main Objective:

To evaluate the association between motor skills and sensory processing in children aged 4 to 11 years with either typical or atypical neurodevelopment (e.g., ASD, ADHD, and DCD).

Secondary Objectives:

To describe and compare motor skills among children aged 4 to 11 years with typical or atypical neurodevelopment, such as ASD, ADHD, and DCD.

To describe and compare sensory processing among children aged 4 to 11 years with typical or atypical neurodevelopment, such as ASD, ADHD, and DCD.

Methodology The study is a cross-sectional observational case-control study. Participants are users of the Child Development and Early Intervention Center (CDIAP) Tris Tras, Neuro Xics, or Criv in Vic.

The sample will include 30 children as controls (typical neurodevelopment) and 10 children as cases (atypical neurodevelopment: ASD, ADHD, DCD).

Children will be assessed using the Infant Motor Profile (IMP) to measure motor development and the Short Sensory Profile-2 (SSP-2) to evaluate sensory processing.

Statistical Analysis Quantitative variables will be described using means and standard deviations, while categorical variables will be presented as frequencies and percentages. Statistical tests such as the Student's t-test will be used to compare means between two groups, ANOVA for comparisons among more than two groups, and the Chi-square test to analyze associations between categorical variables.

Expected Results The study is expected to provide essential insights into the differences in motor development between children with typical and atypical neurodevelopment, as well as the relationship between biological and external factors and these differences. These findings could help improve clinical and educational interventions for these children by tailoring them to their specific needs, thereby enhancing their overall well-being and development.

Ethical Considerations The study protocol will be submitted to the Research Ethics Committee (CER) of UVic-UCC, adhering to good clinical practice guidelines in accordance with the Declaration of Helsinki. Participants will be assigned a code to ensure data pseudonymization, with data securely stored on the Microsoft 365 server of UVic-UCC. Participants will have the right to withdraw from the study at any time, and personal data will be deleted once the study is completed.

Researchers will ensure confidentiality as dictated by Organic Law 3/2018 of December 5 on the Protection of Personal Data and Guarantee of Digital Rights, Regulation (EU) 2016/679 of April 27, 2016, on data protection, and complementary regulations, as well as Organic Law 1/1982 of May 5 on the right to honor, personal and family privacy, and self-image.

DETAILED DESCRIPTION:
Methodology Study Design This study is a cross-sectional observational case-control study designed to generate hypotheses.

The STROBE guidelines will be followed to ensure methodological rigor and transparency in reporting results.

Study Population and Setting The cohort will include children aged 4 to 11 years with typical or atypical neurodevelopment (ASD, ADHD, or DCD).

Participants

Inclusion Criteria:

Children aged 4 to 11 years.

Typical or atypical neurodevelopment, defined as follows:

ASD: Subclinical symptoms or Level 1 diagnosis. ADHD: Predominantly inattentive, hyperactive/impulsive, or combined presentation. For children under 6, typical symptoms of the disorder (e.g., impulsivity, hyperactivity).

DCD: Diagnosed or meeting the following criteria:

Motor skills below age expectations. Significant impact on daily activities or school performance. Difficulties not attributable to another condition. Parental/legal guardian consent.

Exclusion Criteria:

Moderate to severe intellectual disability (IQ ≤ 51). Neurological disorders (e.g., cerebral palsy) or syndromes. Severe visual and/or auditory impairments. Severe behavioral disorders. Severe mental health disorders (e.g., depression, severe anxiety). Participant Recruitment Recruitment will occur between September and October 2024.

Atypical neurodevelopment cases will be recruited from CDIAP Tris Tras, Neuro Xics, and Criv, with service coordinators pre-informed and trained in study procedures and eligibility criteria. Coordinators will review criteria among their clients, provide study details to parents/legal guardians, and share an information sheet and video link explaining the project.

Typical neurodevelopment controls will be recruited from the local community around the research team. Recruitment will follow the same procedure as for atypical cases.

Parents/legal guardians will have 2-5 days to review the study details and sign an informed consent form via Microsoft 365 Forms, ensuring secure data collection.

Sample Size Due to the exploratory nature of this undergraduate project and resource constraints, a formal sample size calculation was not performed. The target is 15 controls (typical neurodevelopment) and 15 cases (5 each for ASD, ADHD, and DCD). This sample size is expected to provide a basis for exploring group-specific dynamics and patterns for future studies.

Variables and Data Collection Independent Variables

Parental Demographics: Age, education level, origin, number of children. Child Demographics: Age, gestational age, birth weight, family type, development type (typical/atypical with diagnosis).

Dependent Variables

Primary Variable:

Motor skills, assessed using the Movement Assessment Battery for Children-Second Edition (MABC-2). This standardized tool evaluates manual dexterity, coordination, and balance through age-adjusted scores. Evaluations will be video-recorded for consistency and scored by trained researchers.

Secondary Variable:

Sensory processing, assessed using the Short Sensory Profile-2 (SSP-2), a caregiver-reported questionnaire evaluating sensory patterns across various domains.

Statistical Analysis Descriptive statistics will summarize quantitative variables using means/standard deviations and medians/interquartile ranges. Categorical variables will be reported as frequencies and percentages. Baseline comparisons will use Student's t-tests or ANOVA for quantitative variables and Chi-square tests for categorical data.

Multivariate analyses will use mixed-effects linear models to evaluate primary outcomes, controlling for significant covariates. Statistical significance is set at p < 0.05.

Ethical Considerations The protocol was approved by the UVic-UCC Research Ethics Committee. The study complies with the Declaration of Helsinki and data protection laws (GDPR and Spanish Organic Law 3/2018).

Parents/legal guardians will receive information sheets and sign informed consent forms. Participation is voluntary, and participants can withdraw at any time without consequences. Video recordings will be securely stored and used solely for study purposes, with images anonymized and deleted after evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 to 11 years.
* Typical or atypical neurodevelopment, defined as follows:
* ASD: Subclinical symptoms or Level 1 diagnosis.
* ADHD: Predominantly inattentive, hyperactive/impulsive, or combined presentation. For children under 6, typical symptoms of the disorder (e.g., impulsivity, hyperactivity).
* DCD: Diagnosed or meeting the following criteria:

  * Motor skills below age expectations.
  * Significant impact on daily activities or school performance.
  * Difficulties not attributable to another condition.
* Parental/legal guardian consent.

Exclusion Criteria:

* Moderate to severe intellectual disability (IQ ≤ 51).
* Neurological disorders (e.g., cerebral palsy) or syndromes.
* Severe visual and/or auditory impairments.
* Severe behavioral disorders.
* Severe mental health disorders (e.g., depression, severe anxiety).

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The cohort will include children aged 4 to 11 years with typical or atypical neurodevelopment (ASD, ADHD, or DCD). Participants will be recruited from the Child Development and Early Intervention Center (CDIAP) Tris Tras, Neuro Xics, and Criv in Vic.
  CDIAP is a free service integrated into the social services network managed by Fundació Sant Tomàs, a non-profit organization in the Osona region.
  Neuro Xics and Criv are private services for child neurodevelopment. Participants with atypical neurodevelopment (ASD, ADHD, or DCD) will be considered cases, while those with typical neurodevelopment will be controls.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Development of Motor Skills | from enrollment to 1 month
  Conducted using the Movement Assessment Battery for Children-Second Edition (MABC-2). This is an internationally recognized standard assessment tool widely used to evaluate motor skills in children aged 4 to 16 years. Consists of three main subtests: Manual Dexterity: evaluates the precision of manual movements and hand-eye coordination through activities such as dragging and releasing objects, drawing straight lines, and working with puzzle pieces.
  Body Coordination: assesses general body coordination and movement planning through activities such as jumping along a line, bouncing a ball, and walking heel-to-toe.
  Balance: evaluates the child's ability to maintain balance in various situations, such as walking on a narrow surface, jumping rope, and standing on one foot for a specified time.
  Standardized scores are provided based on the child's age. Higher score means a better motor skills. Score will be translate to percentile.

SECONDARY OUTCOMES:
Sensory processing | From recruitment to 1 month
  Sensory processing will be assessed using the Short Sensory Profile-2 (SSP-2), a tool designed to evaluate sensory patterns in children aged 3 to 14 years.
  The SSP-2 consists of 38 items that assess various sensory domains (tone modulation, oral sensory response, visuomotor coordination, auditory discrimination, visual perception, and sensory reactivity). Each item is presented as a statement, and parents or guardians rate the frequency with which the child exhibits each behavior on a 5-point scale ranging from "never" to "always." Completing the questionnaire will take approximately 15 minutes. During this time, an experienced occupational therapist will be available to address any.
  Higher raw scores indicate more frequent behaviors related to sensory processing, and lower raw scores represent less frequent behaviors. The raw scores will be converted into standardized values.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vic - Central University of Catalonia, Vic, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly to ensure the confidentiality and privacy of the participants, as outlined in ethical guidelines and legal regulations, including the General Data Protection Regulation (GDPR) and Spanish Organic Law 3/2018 on Data Protection and Guarantee of Digital Rights. Sharing IPD could pose risks of re-identification, especially in a small sample size with specific demographic and clinical characteristics.
  Additionally, this study involves sensitive data related to children and their developmental profiles, requiring strict adherence to data protection standards. Any access to data will be limited to authorized researchers and regulatory bodies as specified in the informed consent, ensuring data use solely for the intended purposes of this study. Aggregate or anonymized results may be shared in publications or presentations to advance knowledge while maintaining participant anonymity.

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/17541055/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/22171930/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/17994185/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/7684363/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/22940157/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/16712636/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/18615927/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/14624826/